CLINICAL TRIAL: NCT06894472
Title: A Comparative Study of EMG Biofeedback and Pharmacotherapy for the Treatment of Masticatory Muscle Hyperactivity in Bruxism Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdullah mohamed elsamahy, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPTBSUREC/0805/2325
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromyography biofeedback + Pharmacotherapy (Experimental): This group will be treated with electromyography biofeedback for one month with a frequency of 3 sessions/week in addition to the pharmacotherapy which prescribed by the dentist.
  Interventions: Other: Electromyography biofeedback; Drug: Pharmacotherapy
- Pharmacotherapy (Other): This group will be treated only with the pharmacotherapy which prescribed by the dentist.
  Interventions: Drug: Pharmacotherapy

INTERVENTIONS:
Other: Electromyography biofeedback — Participants in the experimental group will receive surface electromyography (SEMG) feedback training, targeting the Masseter muscle, for 40 minutes per session according to the Evidence-Based practice since longer practice may become counterproductive due to fatigue and loss of focus. The frequency of the sessions will be 3 sessions/week for 4 weeks.
  Arms: Electromyography biofeedback + Pharmacotherapy
Drug: Pharmacotherapy — Pharmacotherapy will be received by all participants in the two groups in the form of multi relaxant (cyclobenzaprine) 10 MG twice daily for 4 weeks & anti inflammatory (non steroidal anti-inflammatory drugs).

SUMMARY:
This study examines the effect of electromyography biofeedback on masticatory muscles hyperactivity on patients with bruxism.

DETAILED DESCRIPTION:
Bruxism is a movement disorder characterized by excessive activity of the masticatory muscles, resulting in teeth clenching and grinding. It affects 50% to 95% of the adult population. Unlike normal, voluntary chewing movements associated with eating, bruxism involves involuntary jaw muscle contractions that cause tension, leading to muscle soreness and pain. Common symptoms include localized muscle tenderness, orofacial pain, anxiety, stress, fatigue, headaches (especially in the temporal region), restricted mouth opening, and temporomandibular joint stiffness. These symptoms can disrupt sleep, causing transitions from deep to light sleep, increased micro-arousals, and sleep fragmentation, leading to daytime fatigue that impacts social life and work performance.

Bruxism can also lead to masticatory muscle hypertrophy (especially the masseter), tongue burning, linea alba on the cheeks, excessive tooth wear, damage to dental prosthetics, changes in saliva secretion, severe craniofacial pain, and TMJ stiffness. Common treatments for bruxism-related pain often involve medications like Botox, clonazepam, or diazepam, but these are typically temporary and do not address the underlying causes. Moreover, long-term use of these medications may cause complications, and their high cost can limit accessibility.

Non-pharmacological treatments for bruxism include biofeedback, muscle relaxation exercises, occlusal splint therapy, and psychotherapy. Biofeedback, which provides real-time information on bodily functions, helps individuals recognize and modify harmful behaviors. Electromyography (EMG) biofeedback, recognized as effective for temporomandibular disorders (including bruxism), is endorsed by the American Association of Psychophysiology and Biofeedback (AAPB) as an evidence-based intervention.

This study aims to compare the effects of EMG biofeedback training versus oral medications in reducing masticatory muscle hyperactivity in bruxism patients, focusing on addressing the underlying pathophysiology, a topic that, to the authors' knowledge, has not been explored in previous research.

ELIGIBILITY:
Inclusion Criteria:

* Twenty adult subjects with definite mild to moderate bruxism examined by a dentist prior to the study.
* Tenderness of masticatory muscles on palpation grade one and two according to the digital palpating scale
* Mild to moderate myofascial pain around the temporomandibular joint causing discomfort in the morning.

Exclusion Criteria:

* Took any Botox or PRP injection treatment for this condition for the last six months
* Had any advanced periodontal disease.
* Any intraoral fixed splints.
* Pregnancy.
* Under psychiatric care.
* Parkinson
* Have any visual or auditory impairment.
* Any cervical posture abnormalities.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-26 (Estimated); Primary Completion 2025-04-26 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Masseter Hyperactivity | 4 weeks
  The assessment of Masseter muscle hyperactivity will be carried out by the digital palpating scale according to the following criteria: Grade Zero (0): when the muscle palpated and there is no pain or tenderness reported by the patient. Grade (1): Recorded if the patient response the palpation is uncomfortable (tenderness or soreness). Grade (2): is recorded if the patient experiences definite discomfort or pain. Grade (3): is recorded if the patient shows evasive action or eye tearing or verbalizes a desire not to have the area palpated again.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Abdullah mohamed elsamahy, PhD, Principal Investigator — Lecturer; Mohamed Farouk Abdel-Latif, PhD, Principal Investigator — Lecturer; Amal Ahmed Mohamed Morsi, PhD, Principal Investigator — Lecturer; Wafaa Atef Abd Allah, PhD, Principal Investigator — Lecturer; Myassar Ayman Amine, M.Sc, Principal Investigator — Ass. Lecturer
Locations (1):
- Misr University for Science and Technology, Giza, Egypt